CLINICAL TRIAL: NCT03621891
Title: Alterations in Subgingival Microbiota and Hypoxia in Occlusal Trauma
Status: Completed | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Hatice Balci Yuce, Dr, principal investigator, Tokat Gaziosmanpasa University
Other Study IDs: balciyuce84
Record Dates: First submitted 2018-08-04; First posted 2018-08-09 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Chronic Periodontitis; Occlusal Trauma
Keywords: hyper-occlusion; hypoxia; occlusal trauma; periodontitis; subgingival microbiota
MeSH Terms: conditions — Chronic Periodontitis; Hypoxia; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy individuals: Orally and systemically healthy individuals who has no hypo-functional teeth, hyper-occlusion or occlusal trauma
- periodontitis patients: Systemically healthy individuals who has chronic periodontitis but no hypo-functional teeth, hyper-occlusion or occlusal trauma
- healthy-occlusal trauma: Orally and systemically healthy individuals who has occlusal trauma caused by bruxism
- periodontitis-occlusal trauma: Systemically healthy individuals who has both chronic periodontitis and occlusal trauma caused by bruxism

SUMMARY:
Present study suggests that excessive occlusal forces did not cause a significant change in hypoxia and vascular markers, however a slight alteration in subgingival microbiota was observed.

DETAILED DESCRIPTION:
Occlusal trauma is defined as tissue destruction and/or injury resulting in tissue changes in the periodontium as a consequence of excessive occlusal forces or hyper-occlusion. Previous studies suggested accelerated periodontal destruction around teeth with occlusal trauma and increased mobility, however, the evidence is lacking. Recent animal studies found that occlusal trauma increased osteoclastic activity and alveolar bone loss. One possible mechanism suggested for the progression of periodontal destruction with occlusal trauma is that tooth mobility creates a subgingival environment conducive to overgrowth by periodontal pathogens. However, the association of occlusal trauma and subgingival microbiota was not evaluated in previous studies. Therefore, present study aimed to evaluate subgingival dental plaque components and compare with healthy individuals and periodontitis patients without occlusal trauma.

ELIGIBILITY:
Inclusion Criteria:

* Systemical health
* No drug use
* No pregnancy or lactation For group 3 and 4;
* Bruxism at least for 2 years
* Occlusal trauma
* Existence of at least 20 functioning teeth

Exclusion Criteria:

* Smoking
* Pregnancy/lactation
* Systemical disease
* Drug use
* Absence of at least 20 functioning teeth

Ages: 29 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of 80 participants and 4 study groups were created as follows:
  Group 1; healthy individuals without occlusal trauma (Group 1, n=20), 6 men and 14 women, mean age 32.06±2.90 Group 2; periodontitis patients without occlusal trauma (Group 2, n=20), 6 men and 14 women, mean age 36.90±4.67 Group 3; healthy individuals with occlusal trauma (Group 3, n=20), 5 men and 15 women, mean age 34.89±7.51 Group 4; periodontitis patients with occlusal trauma (Group 4, n=20) 7 men and 13 women, mean age 36.76±4.40.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Determination of certain bacterial species in subgingival dental plaque | A day after initial examination
  Subgingival dental plaque samples were collected from each participant and evaluated via polymerase-chain reaction.

SECONDARY OUTCOMES:
hypoxic changes in gingiva and serum | One day after initial examination
  Determination of the hypoxia inducible factor-alpha and vascular endothelial growth factor via ELISA

CONTACTS AND LOCATIONS:
Overall Officials: HATICE BALCI YUCE, PhD, Principal Investigator — Gaziosmanpasa University
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziosmanpasa University Faculty of Dentistry, Tokat Province
  - Gaziosmanpasa University, Tokat Province

IPD SHARING:
Plan to Share IPD: Undecided